CLINICAL TRIAL: NCT03789214
Title: Medical Management of Sleep Disturbance During Opioid Tapering
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00198426; UG3DA048734 (NIH)
Record Dates: First submitted 2018-12-26; First posted 2018-12-28 (Actual); Results first posted 2022-08-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-07

CONDITIONS: Opioid Dependence; Opioid Withdrawal; Sleep Disturbance
MeSH Terms: conditions — Opioid-Related Disorders; Parasomnias | interventions — suvorexant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo sleep medication (Placebo oral capsule)
  Interventions: Drug: Placebo oral capsule
- Low Dose Suvorexant (Active Comparator): Low dose sleep medication
  Interventions: Drug: Low Dose Suvorexant
- High Dose Suvorexant (Active Comparator): High dose sleep medication
  Interventions: Drug: High Dose Suvorexant

INTERVENTIONS:
Drug: Placebo oral capsule — Placebo Sleep Medication
  Arms: Placebo
Drug: Low Dose Suvorexant — Low Dose Suvorexant
  Arms: Low Dose Suvorexant
Drug: High Dose Suvorexant — High Dose Suvorexant
  Arms: High Dose Suvorexant

SUMMARY:
This study will evaluate whether a dual orexin-receptor antagonist approved by the FDA for sleep disturbance, suvorexant (SUVO; Belsomra), will increase total sleep time in patients with opioid use disorder (OUD) undergoing supervised withdrawal. This study is designed as a dose-finding study of SUVO compared to placebo. Briefly, OUD patients seeking supervised withdrawal will be admitted into a clinical research unit and stabilized onto buprenorphine for three days before being randomly assigned to study condition. All participants will then undergo a routine four-day buprenorphine taper, followed by a four-day post-taper phase. Participants will be randomized to receive either placebo, Low Dose SUVO, or High Dose SUVO and the investigators hypothesize that one or both doses of SUVO will improve total sleep time relative to placebo. Patients will attend a single follow-up session, 5-10 days following discharge.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years old and above
* Meets Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 criteria for OUD with evidence of physical dependence on opioids, and seeking treatment to stop using illicit opioids.
* Provides a urine sample that tests positive for opioids.
* Willing to comply with the study protocol.
* Have no clinically significant chronic medical or surgical disorders or conditions that are judged by the investigators to prevent participation.

Exclusion Criteria:

* Seeking or currently enrolled in methadone or buprenorphine maintenance treatment for OUD
* Pregnant or breast feeding
* Have evidence of physical dependence on alcohol or benzodiazepines that requires medical detoxification
* Have a known allergy to the study medications
* Past 30-day prescribed use of suvorexant or benzodiazepines for the indication of insomnia
* Current use of a Selective Serotonin Reuptake Inhibitor (SSRI) or Monoamine oxidase (MAO) inhibitor for depression or insomnia, or other medications that are contraindicated with suvorexant
* Current narcolepsy, restless leg syndrome or sleep paralysis
* High risk for current sleep apnea
* Current major depressive disorder
* Past year suicidal behavior
* Severe hepatic or renal impairment

  * Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) >3x ULN
  * Total bilirubin >2x Upper Limit of Normal (ULN)
  * Creatinine >1.5x ULN
* Have circumstances that would interfere with study participation (e.g., impending jail)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-reported male or female
Enrollment: 90 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew S Huhn, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 90 individuals were consented and screened (35 did not meet eligibility criteria), 55 were scheduled for admission (7 did not present for admission), 48 were admitted for buprenorphine induction (2 were found to be ineligible at this stage and another 6 left prior to randomization), 40 were randomized (1 left before receiving study drug and 1 was excluded because of uncontrolled precipitated withdrawal), and 38 were included in the analyses of study outcomes.
Period: Overall Study
Arm/Group | Placebo | Low Dose Suvorexant | High Dose Suvorexant
Started | 12 | 14 | 12
Completed | 8 | 9 | 9
Not Completed | 4 | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Low Dose Suvorexant | High Dose Suvorexant | Total
Number analyzed (Participants) | 12 | 14 | 12 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.0 (10.4) | 36.7 (9.4) | 46.3 (12.7) | 41.1 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 5
  Male | 10 | 13 | 10 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 3 | 8 | 17
  White | 6 | 10 | 4 | 20
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Abuse Liability as Assessed by Visual Analogue Scale
Description: Area-under-the-curve of self-reported feelings of drug "High" on the morning after study drug administration, measured each morning on a 0-100 point visual analogue scale of the question "Last night, did you feel HIGH?". A score of "0" indicates no abuse liability and a score of 100 indicates extreme abuse liability. This will be assessed over four nights during an opioid taper.
Time Frame: 4 nights
Population: Participants who completed the buprenorphine taper. 1 participant dropped out of the high dose suvorexant condition.
Measure: Mean (Standard Deviation); unit: score on a scale*days
Arm/Group | Placebo | Low Dose Suvorexant | High Dose Suvorexant
Number analyzed (Participants) | 12 | 14 | 11
score on a scale*days | 23.9 (33.5) | 20.9 (28.7) | 22.8 (31.0)
Statistical Analysis 1: Comparison: Placebo vs Low Dose Suvorexant vs High Dose Suvorexant; Test type: Other — One-way ANOVA; p = .950, ANOVA

2. Primary Outcome: Total Sleep Time During Buprenorphine Taper
Description: Area-under-the-curve scores of total number of minutes slept per night as measured by a 3-lead wireless electroencephalography and wrist worn actigraphy.
Time Frame: Four nights during a buprenorphine taper
Population: Participants who completed the buprenorphine taper. 1 participant dropped out of the high dose suvorexant condition.
Measure: Mean (Standard Deviation); unit: minutes*nights
Arm/Group | Placebo | Low Dose Suvorexant | High Dose Suvorexant
Number analyzed (Participants) | 12 | 14 | 11
minutes*nights | 891.6 (287.9) | 1183.6 (300.1) | 1098.4 (287.3)
Statistical Analysis 1: Comparison: Placebo vs Low Dose Suvorexant vs High Dose Suvorexant; Test type: Other — One-way ANOVA; p = .048, ANOVA

3. Primary Outcome: Total Sleep Time During Post-taper
Description: as for outcome 2
Time Frame: Four nights following buprenorphine discontinuation
Population: Prior to completion of the post-taper phase, 4 participants dropped out from the placebo condition, 5 dropped out from the low-dose suvorexant condition, and 3 dropped out from the high-dose suvorexant condition.
Measure: Mean (Standard Deviation); unit: minutes*nights
Arm/Group | Placebo | Low Dose Suvorexant | High Dose Suvorexant
Number analyzed (Participants) | 8 | 9 | 9
minutes*nights | 1049.3 (253.6) | 1113.2 (342.1) | 1055.9 (274.5)
Statistical Analysis 1: Comparison: Placebo vs Low Dose Suvorexant vs High Dose Suvorexant; Test type: Other — One-way ANOVA; p = .691, ANOVA

4. Primary Outcome: Subjective Opiate Withdrawal Scale During Buprenorphine Taper
Description: Area-under-the-curve of peak daily scores on the Subjective Opiate Withdrawal Scale (SOWS) (a 16-item self-reported scale that measures individual opioid withdrawal symptoms using a 0-4 Likert scale; total range of SOWS is 0-64; lower scores indicate mild opioid withdrawal relative to higher scores which indicate more severe opioid withdrawal).
Time Frame: Three days during a buprenorphine taper
Population: Participants who completed the buprenorphine taper. 1 participant dropped out of the high dose suvorexant condition.
Measure: Mean (Standard Deviation); unit: score on a scale*days
Arm/Group | Placebo | Low Dose Suvorexant | High Dose Suvorexant
Number analyzed (Participants) | 12 | 14 | 11
score on a scale*days | 15.5 (12.0) | 10.8 (15.1) | 14.8 (11.2)
Statistical Analysis 1: Comparison: Placebo vs Low Dose Suvorexant vs High Dose Suvorexant; Test type: Other — One-way ANOVA; p = .620, ANOVA

5. Primary Outcome: Subjective Opiate Withdrawal Scale During Post-taper
Description: as for outcome 4
Time Frame: Three days following buprenorphine discontinuation
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale*days
Arm/Group | Placebo | Low Dose Suvorexant | High Dose Suvorexant
Number analyzed (Participants) | 8 | 9 | 9
score on a scale*days | 17.9 (15.1) | 9.0 (9.8) | 6.4 (3.9)
Statistical Analysis 1: Comparison: Placebo vs Low Dose Suvorexant vs High Dose Suvorexant; Test type: Other — One-way ANOVA; p = .067, ANOVA

ADVERSE EVENTS:
Time Frame: 11 days of residential treatment and 5-10 days of follow-up (16-21 days total).
Description: Adverse events represent all events rated as "possibly, probably, or definitely" related to study participation before and after study drug (suvorexant or placebo) administration. All participants received buprenorphine/naloxone for three days prior to randomization, and adverse events in this section may represent events that occurred prior to study drug administration but within the 11 day experimental period because some events persisted across study phases.
Groups:
- Pre-randomization: Pre-randomization to Suvorexant or placebo groups
Arm/Group | Placebo | Low Dose Suvorexant | High Dose Suvorexant | Pre-randomization
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/14 | 0/12 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/14 | 0/12 | 0/38
Other Adverse Events (participants affected / at risk) | 6/12 | 8/14 | 7/12 | 10/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=12) | Low Dose Suvorexant (N=14) | High Dose Suvorexant (N=12) | Pre-randomization (N=38)
Headache (General disorders) | 6 | 3 | 2 | 5 — Headache
Abdominal Cramp (Gastrointestinal disorders) | 1 | 0 | 0 | 3
Abdominal Distention (Gastrointestinal disorders) | 3 | 0 | 1 | 4
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 2 | 1 | 2
Indigestion (Gastrointestinal disorders) | 1 | 0 | 0 | 4
Prolonged Erection (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 — Did not meet criteria for priapism
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 1
Confusion (Nervous system disorders) | 0 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Dream Abnormal (Nervous system disorders) | 4 | 2 | 3 | 0
Drowsiness (Nervous system disorders) | 1 | 1 | 2 | 1
Euphoria (Nervous system disorders) | 1 | 2 | 0 | 0
Impaired/Groggy (Nervous system disorders) | 1 | 2 | 0 | 0
Hypertension (Cardiac disorders) | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Appetite Decreased (General disorders) | 0 | 0 | 0 | 1
Appetite Increased (General disorders) | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Dyspensia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Flatulance (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain Lower Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Insomnia (Nervous system disorders) | 1 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 1 | 0 | 0 | 0
Light headed (Nervous system disorders) | 1 | 0 | 0 | 2
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0
Stuttering/Fluency Disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Photophobia (Eye disorders) | 1 | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Sweat Increased (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Blurred Vision (Eye disorders) | 1 | 0 | 0 | 0
Itchy Eyes (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Eye Pain (Eye disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-04): https://cdn.clinicaltrials.gov/large-docs/14/NCT03789214/Prot_SAP_002.pdf
  • Informed Consent Form (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/14/NCT03789214/ICF_001.pdf